CLINICAL TRIAL: NCT04820855
Title: Mindfulness and Yoga for Pain With Interstitial Cystitis Evaluation
Acronym: MYPAICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-664
Record Dates: First submitted 2021-03-15; First posted 2021-03-29 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial cystitis; Complementary and Alternative medicine; Yoga; Meditation
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Therapeutics; Mind-Body Therapies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): This is an individual treatment program devised by a pelvic floor physical therapist including a daily yoga series and mindfulness via a Smartphone app.
  Interventions: Behavioral: Treatment; Other: Usual Cares
- Control (Active Comparator): These are participants undergoing regular treatment for interstitial cystitis with their providers
  Interventions: Other: Usual Cares

INTERVENTIONS:
Behavioral: Treatment — This is the treatment program devised win conjunction with a pelvic floor physical therapist. It is a daily yoga series and mindfulness with a Smartphone app.
  Other Names: Mind/Body Therapy
  Arms: Treatment
Other: Usual Cares — This is standard treatment for Interstitial cystitis with your provider.
  Other Names: Standard Cares

SUMMARY:
This study is examining impact of pain on daily life, the ability to function and treatments used for patients with interstitial cystitis/painful bladder syndrome before and after a program of mindfulness and yoga, in comparison to patients who are undergoing treatment with their providers.

DETAILED DESCRIPTION:
This is a randomized control trial comparing women diagnosed with interstitial cystitis/painful bladder syndrome (ICPBS) receiving usual ICPBS care to those treated with usual care supplemented with meditation and yoga. Both groups continued their current ICPBS treatment regimens. Participants in the intervention group additionally received a commercially available meditation application and a yoga tutorial video. Women in either group were followed weekly for three months. Validated questionnaires were used to compare treatment response from baseline to 12 weeks of intervention for both groups. The primary outcome was the patient report on the global response assessment (GRA), and we required a sample size of 82 patients (41 per group) to detect a difference of 30% with a 10% margin of error (alpha of 0.05) with 80% power. Other questionnaires collected included the PROMIS pain interference scale, the interstitial cystitis problem index and symptom index (ICPI and ICSI), the VAS pain scale, treatment compliance, and treatment escalation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* >=Age 18
* IC/BPS diagnosis
* English or Spanish reading/writing
* Own a Smartphone and able to watch online yoga tutorials
* Ability/willingness to participate in follow up questionnaires
* ICSI/ICPI >6 at baseline
* Physical exam in the past 2 years by urogynecology or gynecologist

Exclusion Criteria:

* Pregnancy or lactating
* Inability to speak/write in English/Spanish
* Known history of recurrent UTI
* Urinary retention ( PVR>150 ml)
* History of augmentation cystoplasty or urinary diversion.
* History of chemotherapy/radiation or radiation induced cystitis
* Hunner's Ulcers demonstrated in last 6 months by cystoscopy
* Parkinsonism with neurogenic bladder
* Multiple Sclerosis with neurogenic bladder
* CVA with residual deficits
* Patients with severe mobility impairment and inability to perform yoga postures
* Patients who are hard of hearing or visually impaired
* Imprisoned patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Meriwether, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dao AN, Komesu YM, Jansen SM, Petersen TR, Meriwether KV. Augmentation of Interstitial Cystitis-Bladder Pain Syndrome Treatment With Meditation and Yoga: A Randomized Controlled Trial. Obstet Gynecol. 2025 Feb 1;145(2):186-195. doi: 10.1097/AOG.0000000000005820. Epub 2025 Jan 2. PMID 39746210

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 49 | 48
Completed | 43 | 39
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (15) | 50 (17) | 49.3 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 46 | 44 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97
Education [Number; unit: participants]
  HIgh schooil or high school equivalency certificate | 9 | 7 | 16
  Associate degree | 9 | 8 | 17
  4y college degree | 19 | 15 | 34
  Graduate degree | 12 | 17 | 29
  Unknown or not recorded | 0 | 1 | 1
Marital status [Number; unit: participants]
  Single | 10 | 12 | 22
  Married | 28 | 25 | 53
  Divorced, separated, widowed | 11 | 11 | 22
History of substance use disorder [Number; unit: participants] | 3 | 2 | 5
Age of diagnosis of ICBPS [Median (Inter-Quartile Range); unit: years] | 45 [27 to 53] | 39 [28 to 52] | 41.2 [25 to 57]
Interstitial Cystitis Symptom Index Score [Mean (Standard Deviation); unit: units on a scale] — The Interstitial Cystitis Symptoms Index Scale (ICSI) is a scale of point ranging from 0 to 20, with higher scores indicating WORSE OUTCOMES (more symptoms)
  units on a scale | 11.7 (3.6) | 13.2 (4.4) | 12.4 (4.1)
Interstitial Cystitis Problem Index Score [Mean (Standard Deviation); unit: units on a scale] — The Interstitial Cystitis Problem Index Scale (ICPI) is a scale of point ranging from 0 to 16, with higher scores indicating WORSE OUTCOMES (more problems)
  units on a scale | 10 (3.2) | 11.2 (3.3) | 10.6 (3.3)
Pain Visual Analog Scale Score [Mean (Standard Deviation); unit: units on a scale] — The Pain Visual Analog Scale (VAS) Score ranges from 1 to 10, with patients ranking their pain from no pain (score of 0) to most severe pain imaginable (score of 10), with high scores indicating WORSE OUTCOMES (more pain)
  units on a scale | 4.8 (2.3) | 5.0 (2.1) | 4.9 (2.2)
Hospital Anxiety and Depression anxiety score [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS) anxiety subscale has a score range from 0 to 21, with higher scores indicating greater anxiety levels (WORSE OUTCOMES). Each item on the scale is scored from 0 to 3, contributing to the total possible score of 21 for the anxiety subscale at most (highest level of anxiety).
  A score of 0-7 is generally considered normal, 8-10 as mild anxiety, 11-14 as moderate anxiety, and 15 or higher as severe anxiety.
  units on a scale | 9.7 (3.9) | 9.1 (4.3) | 9.4 (4.1)
Hospital Anxiety and Depression depression score [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS) depression subscale has a score ranging 0 to 21, with higher scores indicating greater levels of depression (WORSE OUTCOME). Each item on the scale is scored from 0 to 3, contributing to the total possible score of 21 for the depression subscale at most (highest level of depression).
  units on a scale | 5.3 (3.6) | 6.3 (4.3) | 5.8 (4.0)
PROMIS Pain Interference Score [Mean (Standard Deviation); unit: units on a scale] — The PROMIS Pain Interference Scale (PIS) has a raw score ranging from 5 to 30, with higher scores indicating a greater level of pain interference in life (WORSE OUTCOMES).
  units on a scale | 17.5 (5.6) | 18.3 (6.0) | 17.9 (5.8)
Pain self efficacy score [Mean (Standard Deviation); unit: units on a scale] — The Pain Self-Efficacy Questionnaire (PSEQ) score ranges from 0 to 60, with higher scores indicating a greater belief in one's ability to manage pain and function (BETTER OUTCOMES).
  units on a scale | 7.1 (2.5) | 7.2 (2.4) | 7.15 (2.4)
Prior treatments [Number; unit: participants]
  Education, behavioral modification, stress management | 23 | 21 | 44
  Medications, intravesical instillations, physical therapy | 48 | 48 | 96
  Cystoscopic hydrodistension under general anesthesia | 2 | 3 | 5
  Intradetrusor botulinum toxin A, sacral neuromodulation | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Designated as "Treatment Responders" Based on Global Response Assessment (GRA)
Description: This is a validated single question that determines treatment response. Participants were considered "treatment responders" if they answered "markedly improved/moderately improved" on the GRA at 12 weeks.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
Participants | 31 | 10

2. Secondary Outcome: O'Leary-Sant: Interstitial Cystitis Symptom Index
Description: This is a validated questionnaire to evaluate interstitial cystitis symptoms. The Interstitial Cystitis Symptoms Index Scale (ICSI) is a scale of point ranging from 0 to 20, with higher scores indicating WORSE OUTCOMES (more symptoms)
Time Frame: change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
score on a scale | -3.4 (3.7) | -1.5 (3.9)

3. Secondary Outcome: O'Leary-Sant: Interstitial Cystitis Problem Index
Description: The Interstitial Cystitis Problem Index Scale (ICPI) is a scale of point ranging from 0 to 16, with higher scores indicating WORSE OUTCOMES (more problems)
Time Frame: change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
score on a scale | -3.7 (3.2) | -1.9 (2.8)

4. Secondary Outcome: Pain VAS Score
Description: The Pain Visual Analog Scale (VAS) Score ranges from 1 to 10, with patients ranking their pain from no pain (score of 0) to most severe pain imaginable (score of 10), with high scores indicating WORSE OUTCOMES (more pain)
Time Frame: change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
score on a scale | -1.7 (2.4) | -0.3 (2.3)

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale
Description: Hospital Anxiety and Depression Scale (HADS) anxiety subscale has a score range from 0 to 21, with higher scores indicating greater anxiety levels (WORSE OUTCOMES). Each item on the scale is scored from 0 to 3, contributing to the total possible score of 21 for the anxiety subscale at most (highest level of anxiety).
  A score of 0-7 is generally considered normal, 8-10 as mild anxiety, 11-14 as moderate anxiety, and 15 or higher as severe anxiety.
Time Frame: change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
score on a scale | -1.6 (2.8) | -0.6 (3.0)

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Depression Subscale
Description: Hospital Anxiety and Depression Scale (HADS) depression subscale has a score ranging 0 to 21, with higher scores indicating greater levels of depression (WORSE OUTCOME). Each item on the scale is scored from 0 to 3, contributing to the total possible score of 21 for the depression subscale at most (highest level of depression).
Time Frame: change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
score on a scale | -1.6 (2.6) | -0.7 (3.3)

7. Secondary Outcome: PROMIS Pain Interference Score
Description: The PROMIS Pain Interference Scale (PIS) has a raw score ranging from 5 to 30, with higher scores indicating a greater level of pain interference in life (WORSE OUTCOMES).
Time Frame: change froom baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
score on a scale | -5.5 (5.9) | -3.1 (6.2)

8. Secondary Outcome: Pain Self-efficacy-2 Score
Description: The Pain Self-Efficacy Questionnaire (PSEQ) score ranges from 0 to 60, with higher scores indicating a greater belief in one's ability to manage pain and function (BETTER OUTCOMES).
Time Frame: change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 43 | 39
score on a scale | 1.5 (3.2) | 0.9 (3.4)

ADVERSE EVENTS:
Time Frame: Over 3 months during study participation.
Description: Participants were contacted weekly during the study period and specifically asked if they experienced any adverse events and data was recorded.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 1/49 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=49) | Control (N=48)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient diagnosed with COVID-19 during course of study; did not require hospitalization or have subsequent sequelae at end of study. Adverse event deemed likely not related to study participation or intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04820855/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT04820855/ICF_001.pdf